CLINICAL TRIAL: NCT03573947
Title: A Phase II Clinical Trial of Combination Nivolumab (Opdivo), Ipilimumab (Yervoy), and Paclitaxel in Patients With Untreated Metastatic Non-Small Cell Lung Cancer (NSCLC) (The OPTIMAL Trial) [TOP 1705]
Brief Title: Phase II Clinical Trial of NIVO-IPI-TAXANE in Untreated Metastatic NSCLC
Acronym: TOP1705
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jeffrey Clarke (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Clarke, Asst. Prof. of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00092210
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Stage IV Non-Small Cell Lung Cancer; nivolumab; ipilimumab; paclitaxel; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- nivolumab, ipilimumab and paclitaxel (Experimental): patients will be treated with nivolumab and ipilimumab in combination with weekly paclitaxel days 1 and 8 every 21 days until they experience unacceptable drug-related toxicity, disease progression or 24 months.
  The dosing regimen will be: nivolumab 360 mg every 3 weeks, ipilimumab 1 mg/kg every 6 weeks, and paclitaxel 80 mg/m2 on days 1 and 8 of 1 21 day treatment cycle. Paclitaxel would be stopped after a total of 4-6 cycles of treatment.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Nivolumab — 360 mg intravenously every 3 weeks
  Other Names: Opdivo
Drug: Ipilimumab — 1 mg/kg intravenously over 30 minutes
  Other Names: Yervoy
Drug: Paclitaxel — 80 mg/m2 on days 1 and 8 of every 21-day treatment cycle
  Other Names: Taxol

SUMMARY:
This is an open-label, non-randomized, phase II clinical research study designed to assess the safety and efficacy of nivolumab and ipilimumab in combination with paclitaxel in patients with treatment naïve NSCLC.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, phase II clinical research study designed to assess the safety and efficacy of nivolumab and ipilimumab in combination with paclitaxel in patients with treatment naïve NSCLC.

Patients with histologically confirmed stage IV or recurrent non curable NSCLC of squamous or non-squamous histology, with no prior systemic anticancer chemotherapy or immunotherapy given as primary treatment for advanced or metastatic disease may be eligible to participate in this study.

Patients enrolled into the study will be given the study drugs, nivolumab (360 mg) (Day 1) every 3 weeks, ipilimumab 1 mg/kg (Day 1) every 6 weeks, and paclitaxel 80mg/m2 on days 1 and 8 of each 21- day study treatment cycle. Paclitaxel will be stopped after a total of 4-6 cycles of treatment. Blood samples and possibly a small piece of tissue may be removed the patient's lung to see what type of lung cancer cells that she or he may have. Patients will also have other tests, exams, and procedures for study purposes and their standard of care. Subject participation in the study will last for up to approximately 48 months after the start of the study drug or until their condition worsens or they experience intolerable adverse events as deemed by the study doctor.

There are possible patient risk to this study that include but are not limited to diarrhea, itching, rash and a feeling of weakness.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage IV or recurrent Non-small cell lung cancer squamous or non-squamous histology (Stage IV as diagnosed using the 7th edition of Lung Cancer Stage Classification), with no prior systemic anticancer therapy given as primary therapy for advanced or metastatic disease. Prior adjuvant chemotherapy, neoadjuvant chemotherapy, or chemoradiotherapy is permitted as long as the last administration of the prior regimen occurred at least 6 months prior to study enrollment. Patients with EGFR, ALK, or ROS1 alterations must have received one prior TKI.
* A core needle biopsy or surgical specimen must be available for submission.
* At least one site of disease that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 that has not been previously irradiated; if the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
* Age ≥ 18 years with ability and willingness to provide informed consent.
* ECOG performance status 0 or 1.
* Negative pregnancy test done ≤72 hours (or per institutional policy) prior to treatment, for women of childbearing potential only. Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  1. Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
  2. Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
  3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* Men and women of childbearing potential must agree to use medically accepted barrier methods of contraception (e.g. male or female condom) at the time of pregnancy test (women of childbearing potential only), during the course of the study and for 90 days after the last dose of study drug, even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of study and for 90 days after the last dose of study drug.
* A concurrent diagnosis of a separate malignancy is allowed if clinically stable and does not require tumor-directed therapy.
* Provision of written informed consent including HIPAA according to institutional guidelines prior to any study-specific procedures
* Patients must agree to research blood sampling to participate in study;
* Adequate organ and marrow function as defined by the following:

  1. Creatinine clearance ≥ 50 cc/min or serum Cr < 1.5 x institutional ULN
  2. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  3. AST/ALT ≤ 2 x ULN without liver metastasis; ≤ 5 x ULN with liver metastasis
  4. Absolute neutrophil count (ANC) ≥ 1500 µl
  5. Hemoglobin (Hgb) ≥ 9 g/dL
  6. Platelets ≥ 100,000/µl

Exclusion Criteria:

* Subjects with known EGFR mutations which are sensitive to available targeted inhibitor therapy and must have received treatment with at least one prior tyrosine kinase inhibitor (TKI).
* Subjects with known ALK or ROS1 translocations which are sensitive to available targeted inhibitor therapy must have received treatment with at least one prior TKI.
* Radiation therapy within 14 days prior to day 1 of study drug.
* Experimental agents within 28 days prior to day 1 of study drug.
* Intolerance of nivolumab or other PD-1/PD-L1 axis drug(s), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including prior therapy with anti-tumor vaccines or other immune-stimulatory anti-tumor agents.
* Known auto-immune conditions requiring systemic immune suppression therapy other than prednisone < 10 mg daily (or equivalent).
* History of interstitial pneumonitis from any cause.
* Concurrent severe and/or uncontrolled medical conditions which may compromise participation in the study, including impaired heart function or clinically significant heart disease.
* Pregnant or breast feeding.
* Not willing to use an effective method of birth control medically accepted barrier methods of contraception (e.g. male or female condom) at the time of pregnancy test (women of childbearing potential only), during the course of the study and for 90 days after the last dose of study drug.
* Current use of medications specified by the protocol as prohibited for administration in combination with the study drugs. This includes patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to day 1 of study drug. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment on day 1 of study drug. Patients receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Known active CNS metastases which are symptomatic. Eligible if metastases have been locally treated 14 days prior to cycle 1 day 1, are clinically controlled, or asymptomatic on cycle 1 day
* Steroid dose must be equivalent of <10 mg prednisone daily or equivalent dose steroid. Untreated, asymptomatic brain metastases allowed if subject does not require corticosteroids or anticonvulsant therapy.
* History of myocardial infarction, NYHA class III or IV congestive heart failure, or unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 6 months prior to study enrollment.
* Known history of HIV seropositivity or known acquired immunodeficiency syndrome (AIDS), hepatitis C virus (allowed if received curative therapy), acute or chronic active hepatitis B infection, or other serious chronic infection requiring ongoing treatment.
* Inability to comply with protocol or study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Clarke, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- nivolumab, ipilimumab and paclitaxel: patients will be treated with nivolumab and ipilimumab in combination with weekly paclitaxel days 1 and 8 every 21 days until they experience unacceptable drug-related toxicity, disease progression or 24 months.
  The dosing regimen will be: nivolumab 360 mg every 3 weeks, ipilimumab 1 mg/kg every 6 weeks, and paclitaxel 80 mg/m2 on days 1 and 8 of 1 21 day treatment cycle. Paclitaxel would be stopped after a total of 4-6 cycles of treatment.
  Nivolumab: 360 mg intravenously every 3 weeks
  Ipilimumab: 1 mg/kg intravenously over 30 minutes
  Paclitaxel: 80 mg/m2 on days 1 and 8 of every 21-day treatment cycle
Period: Overall Study
Arm/Group | nivolumab, ipilimumab and paclitaxel
Started | 46
Completed | 44
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | nivolumab, ipilimumab and paclitaxel
Number analyzed (Participants) | 46
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [61 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46
Smoking status [Count of Participants; unit: Participants]
  Current | 9
  Former | 32
  Never | 5
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 29
  Squamous cell carcinoma | 12
  Adenosquamous | 3
  Large cell with neuroendocrine features | 1
  Mucinous adenocarcinoma | 1
Prior surgery undergone [Count of Participants; unit: Participants]
  Yes | 37
  No | 9
Prior systemic therapy received [Count of Participants; unit: Participants]
  Yes | 5
  No | 41
Prior radiation therapy received [Count of Participants; unit: Participants]
  Yes | 23
  No | 23
Brain metastases at enrollment (yes/no) [Count of Participants; unit: Participants]
  Yes | 14
  No | 32

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Determined by the Investigator Using Response Evaluation Criteria In Solid Tumors RECIST 1.1 (Brand Name) or Death, Whichever Occurs First
Description: Progression-free survival (PFS) will be defined as the time from first dosing date to the date of the first documented tumor progression determined by the investigator using RECIST 1.1 or death, whichever occurs first
Time Frame: up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | nivolumab, ipilimumab and paclitaxel
Number analyzed (Participants) | 46
months | 9.4 [5.9 to 16.6]

2. Secondary Outcome: Description of the Safety and Adverse Events of the Combination Nivolumab, Ipilimumab, and Paclitaxel in Untreated, Metastatic NSCLC.
Description: The study will assess the number and percentage of participants who experience high grade (Grade 3-4 and Grade 5) treatment-related select and immune-mediated adverse events that include: pneumonitis, interstitial nephritis, diarrhea/colitis, hepatitis, rash, endocrinopathies, and hypersensitivity/infusion reaction events.
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | nivolumab, ipilimumab and paclitaxel
Number analyzed (Participants) | 46
Participants
  Fatigue | 24
  Alopecia | 17
  Anorexia | 16
  Infusion-related reaction | 15
  Adrenal insufficiency | 10
  Diarrhea | 10
  Rash maculopapular | 9
  Pneumonitis | 8
  Colitis | 7
  Hypothyroidism | 7

3. Secondary Outcome: Estimate the Overall Response Rate With the Study Combination.
Description: Objective Response Rate (ORR) defined as the number and percentage of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR). Best overall response (BOR) is defined as the best response designation, recorded between the date of first dose and the date of the initial objectively documented tumor progression per RECIST v1.1 or the date of subsequent therapy, whichever occurs first.
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | nivolumab, ipilimumab and paclitaxel
Number analyzed (Participants) | 46
Participants
  Complete response | 2
  Partial response | 20
  Stable disease | 19
  Progressive disease | 5

ADVERSE EVENTS:
Time Frame: up to 4 years
Arm/Group | nivolumab, ipilimumab and paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 26/46
Other Adverse Events (participants affected / at risk) | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | nivolumab, ipilimumab and paclitaxel (N=46)
Adrenal insufficiency (Endocrine disorders) | 5
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Colitis (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Infections and infestations (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Infections and infestations) | 1
Non-cardiac chest pain (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Renal and urinary disorders - Other, Specify (Renal and urinary disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Sepsis (Infections and infestations) | 1
Stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | nivolumab, ipilimumab and paclitaxel (N=46)
Fatigue (General disorders) | 27
Alopecia (Skin and subcutaneous tissue disorders) | 17
Anorexia (Metabolism and nutrition disorders) | 17
Infusion related reaction (General disorders) | 15
Diarrhea (Gastrointestinal disorders) | 11
Adrenal insufficiency (Endocrine disorders) | 9
Hypothyroidism (Endocrine disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Weight loss (Investigations) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Mucosal infection (Infections and infestations) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 4
Hypotension (Vascular disorders) | 4
Lung infection (Infections and infestations) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 3
Atrial fibrillation (Cardiac disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Endocrine disorders - Other, Specify (Endocrine disorders) | 6
Hypertension (Vascular disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Infections and infestations - Other, Specify (Infections and infestations) | 3
Pain (General disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Sinusitis (Infections and infestations) | 3
Thromboembolic event (Vascular disorders) | 3
Thromboembolic event (Infections and infestations) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT03573947/Prot_SAP_000.pdf